CLINICAL TRIAL: NCT03767530
Title: Efficacy and Safety of Thermic Devices in the Treatment of Meibomian Gland Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Collaborators: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Karim Mohamed-Noriega, Professor, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OF18-00006
Record Dates: First submitted 2018-10-31; First posted 2018-12-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-05

CONDITIONS: Meibomian Gland Dysfunction
Keywords: Meibomian gland dysfunction; Mibo; MGD; Dry eye disease; Thermic devices
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: All subjects will be ophthalmologically evaluated before treatment and at weeks 8, 16 and 24. Subjects will be randomly assigned into 2 study groups. Mibo group will have 3 sessions (basal, week 2, week 4) of thermal therapy with Mibo Thermoflo in both eyes. The control group will use warm compresses and eyelid massage 2 times per day in both eyes. At the week 16 control group will also have 3 sessions of Mibo therapy at 2 weeks interval.
Masking Description: Not blinded study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mibo Thermoflo (thermal device) (Experimental): 3 sessions at 2 weeks interval (basal, week 2, week 4)of 11 minutes per eye of thermal therapy with Mibo Thermoflo.
  Interventions: Device: Mibo Thermoflo
- Warm compresses and eyelid massage (Active Comparator): 2 times per day, 11 minutes per eye.
  Interventions: Other: Warm compresses and eyelid massage

INTERVENTIONS:
Device: Mibo Thermoflo — Thermal therapy with Mibo Thermoflo for 11 minutes per eye, during each session.
  Arms: Mibo Thermoflo (thermal device)
Other: Warm compresses and eyelid massage — Warm compresses plus eyelid massage 2 times per day 11 minutes per eye.
  Arms: Warm compresses and eyelid massage

SUMMARY:
Dry eye syndrome is a common eye disease that affects 1 to 2 out of 10 persons around the planet. One common cause of this disease is the meibomian gland dysfunction. Meibomian glands are very small glands located at the rim of the eyelids that produce an oily substance that prevents the evaporation of tears. When these glands are compromised, the tear film evaporates quickly and the eyes dry up. This disease presents as eye irritation, foreign body sensation, inflammation, etc. The treatment of choice for MGD is eyelid massage and warm compresses 2 times a day. However, these treatments not always work perfectly, and as a result, patients find it hard to follow doctor's orders. Another kind of treatment is thermal therapy. There are several devices that are designed to apply heat on the eyelids, such as Lipiflow, MiBo Thermoflo, and Blephasteam. In this study, we want to find out whether thermal therapy with MiBo Thermoflo works better than warm compresses and eyelid massage use in the treatment of dry eye caused by MGD. To do this, we will select several patients and will assign them randomly to either the group with thermal therapy with MiBo Thermoflo or to the group with warm compresses and eyelid massage. The Mibo group will receive 3 sessions of thermal therapy at 2 weeks interval and the control group warm compresses and eyelid massage 2 times per day. All subjects will have a follow up of 24 weeks and we will compare results for both groups at the end of the study.

DETAILED DESCRIPTION:
Dry eye syndrome is considered one of the most important ophthalmologic diseases, affecting 10 to 20% of the general population. Of these, 3.7% to 70% of cases are due to meibomian gland dysfunction (MGD). MGD is a chronic diffuse disease characterized by terminal duct obstruction and/or qualitative/quantitative changes in gland secretion. This causes a disruption in the tear film, ocular irritation symptom, inflammation, and ocular surface symptoms. The gold standard for the treatment of meibomian dysfunction is the use of warm compresses and eyelid massage 2 times a day. These have variable results and consequently patient's adherence to treatment is low. An alternative treatment is the use of thermal therapy devices such as Lipiflow, MiBo Thermoflo, and Blephasteam. The objective of this study is to determine if the thermal device MiBo Thermoflo is more effective than warm compresses and eyelid massage in the treatment of dry eye secondary to MGD. Participants will be randomly assigned to one of two groups: the Mibo group will receive 3 sessions of thermal therapy at 2 weeks interval and the control group warm compresses and eyelid massage 2 times per day. All subjects will have follow up of 24 weeks and we will compare results for both groups at the end of the study. During the protocol patients in both groups will continue with their standard treatment for dry eye as needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with:

  * Dry eye syndrome with meibomian gland dysfunction alone or in combination of other type of dry eye.
  * Patients who were previously treated with eyelid massages and warm compresses without any improvement.

Exclusion Criteria:

* Pregnant women.
* History of ocular surgery within three months prior to inclusion.
* History of trauma, infection or inflammation within three months prior to inclusion.
* Contact lens use in the last week before inclusion.
* Patients with active ocular allergic disease.
* Patient with microbial keratitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Meibomian gland expressibility | Basal to 24 weeks
  Changes in meibomian gland structure will be evaluated by meibomian gland expressibility.
Meibum quality | Basal to 24 weeks
  Changes in meibomian gland structure will be evaluated with the meibum quality in slit lamp graded as: clear, opaque, granular and toothpaste for meibum worst secretion.
Corneal and conjunctival staining with fluorescein dye | Basal to 24 weeks
  Ocular surface damage will be graded with corneal and conjunctival staining with fluorescein dye.
Corneal and conjunctival staining with lissamine green dye | Basal to 24 weeks
  Ocular surface damage will be graded with corneal and conjunctival staining with lissamine green dye.
Tear Break-up Time (TBUT) | Basal to 24 weeks
  Tear stability will be measured with Tear Break-up Time (TBUT). A result >10 seconds will be considered normal, a result <10 seconds will be considered pathological.
Schirmer test with and without anesthesia | Basal to 24 weeks
  Tear production will be measured by Schirmer test with and without anesthesia. A Schirmer test >10 mm will be considered normal, a result >5 mm pathological. The Schirmer test with anesthesia >15 mm is consider normal.
Symptom Assessment in Dry Eye questionnaire (SANDE) | Basal to 24 weeks
  Ocular surface symptoms will be assessed by the Symptom Assessment in Dry Eye (SANDE) questionnaire. The SANDE questionnaire has two questions presented in a visual scale. The two questions assess the frequency and severity of dry eye symptoms.
Ocular Surface Disease Index (OSDI) | Basal to 24 weeks
  Ocular surface symptoms will be assessed by the Ocular Surface Disease Index (OSDI). The OSDI questionnaire consists of 12 questions that assess dry eye symptoms and their effects on vision related function. The questionnaire is divided in 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients are asked to rate their responses on a 0 to 4 scale where 0 represents "none of the time", 1 "some of the time", 2 "half of the time", 3 "most of the time", and 4 "all of the time". The total score is calculated using the following formula: ([sum of scores for all questions answered x 100] / [total number of questions answered x 4]). Lower scores represent a better outcome.
Dry Eye Questionnaire 5 (DEQ-5) | Basal to 24 weeks
  Ocular surface symptoms will be assessed by the Dry Eye Questionnaire 5 (DEQ-5). The Dry Eye Questionnaire 5 asses habitual dry eye symptoms (discomfort, dryness and wetty eyes) and severity level.
Tear osmolarity | Basal to 24 weeks
  Patients with dry eye have increased levels of tear osmolarity wich is one of tear inflammation biomarkers. Tear osmolarity will be performed with Tear Lab Osmolarity System, a result of 308 mOsm/L or higher indicates dry eye disease.
Change in tear of matrix metalloproteinase 9 (MMP-9) | Basal to 24 weeks
  MMP-9 is an inflammatory biomarker wich is elevated in the tears of patients with dry eye and an early diagnostic evaluation, it is realized in consulting room with the InflammaDry test (Rapid Pathogen Screening Inc.). The presence of 1 line is a negative result and two lines means positive result.
Non-Invasive Keratograph Break-up Time (NIKBUT) | Basal to 24 weeks
  NIKBUT will be measured with Keratograph 5M. A JENVIS Dry Eye report will be generated to document findings.
Tear meniscus height | Basal to 24 weeks
  Tear meniscus height will be measured with Keratograph 5M. A JENVIS Dry Eye report will be generated to document findings.
Conjuctival hyperemia | Basal to 24 weeks
  Conjuctival hypermeia will be graded with JENVIS Scale performed by Keratograph 5M. A JENVIS Dry Eye report will be generated to document findings. Conjuctival hyperemia will be . graded as: none, mild moderate or severe.
Lipid layer thickness | Basal to 24 weeks
  Lipid layer thickness will be measured with Keratograph 5M. A JENVIS Dry Eye report will be generated to document findings.
Adverse events | Basal to 24 weeks
  Adverse events will be evaluated during the ophthalmic evaluation.

SECONDARY OUTCOMES:
Short term changes with corneal and conjunctival staining with fluorescein dye | These parameters will be evaluated before sessions of termal therapy at week 2 and week 4
  Short term changes in ocular surface damage will be graded with corneal and conjunctival staining with fluorescein dye.
Short term changes with corneal and conjunctival staining with lissamine green dye | These parameters will be evaluated before sessions of termal therapy at week 2 and week 4
  Short term changes in ocular surface damage will be graded with corneal and conjunctival staining with lissamine green dye.
Short term changes in tear stability | These parameterd will be evaluated before sessions of termal therapy at week 2 and week 4
  Short term changes in tear stability will be measured with Tear Break-up Time (TBUT). A result >10 seconds will be considered normal, a result <10 seconds will be considered pathological.
Short term changes in Symptom Assessment in Dry Eye questionnaire (SANDE) | These parameters will be evaluated before sessions of termal therapy at week 2 and week 4
  Short term changes in ocular surface symptoms will be assessed by the Symptom Assessment in Dry Eye (SANDE). The SANDE questionnaire has two questions presented in a visual scale. The two questions assess the frequency and severity of dry eye symptoms. A less rate prove changes in ocular surface symptoms and quality of life improvement.
Short term changes in Ocular Surface Disease Index (OSDI) | These parameters will be evaluated before sessions of termal therapy at week 2 and week 4
  Short term changes in ocular surface symptoms will be assessed by the Ocular Surface Disease Index (OSDI). The OSDI questionnaire consists of 12 questions that assess dry eye symptoms and their effects on vision related function. The questionnaire is divided in 3 subscales: ocular symptoms, vision-related function, and environmental triggers.. A less rate prove changes in ocular surface symptoms and quality of life improvement.
Short term changes in Dry Eye Questionnaire 5 (DEQ-5) | These parameters will be evaluated before sessions of termal therapy at week 2 and week 4
  Short term changes in ocular surface symptoms will be assessed by the Dry Eye Questionnaire 5 (DEQ-5). The Dry Eye Questionnaire 5 asses habitual dry eye symptoms (discomfort, dryness and wetty eyes) and severity level. A less rate prove changes in coular surface symptoms and quality of life improvement.
Eyelid skin temperature | These parameters will be evaluated before sessions of termal therapy at week 2 and week 4
  Eyelid skin temperature will be measured with the thermographic infrared scientific equipment FLIR SC4000 to verify if 42 celsius degree are obtain as maker recommends.
Corneal conjunctival temperature | These parameters will be evaluated before sessions of termal therapy at week 2 and week 4
  Corneal conjunctival temperature will be measured with the thermographic infrared scientific equipment FLIR SC4000 to verify if 42 celsius degree are obtain as maker recommends.
Bulbar conjunctival temperature | These parameters will be evaluated before sessions of termal therapy at week 2 and week 4
  Bulbar conjunctival temperature will be measured with the thermographic infrrared scientific equipment FLIR SC4000 to verify if 42 celsius degree are obtain as maker recommends.
Tarsal conjunctival temperature | These parameters will be evaluated before sessions of thermal therapy at week 2 and week 4.
  Tarsal conjunctival temperature will be measured with the thermographic infrared scientific equipment FLIR SC4000 to verify if 42 celsius degree are obtain as maker recommends.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Mohamed-Noriega, M.D., Principal Investigator — Departamento de Oftalmologia, Hospital Universitario Dr. Jose Eleuterio Gonzalez
Locations (1):
- Departamento de Oftalmologia, Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arita R, Morishige N, Shirakawa R, Sato Y, Amano S. Effects of Eyelid Warming Devices on Tear Film Parameters in Normal Subjects and Patients with Meibomian Gland Dysfunction. Ocul Surf. 2015 Oct;13(4):321-30. doi: 10.1016/j.jtos.2015.04.005. Epub 2015 May 30. PMID 26031204
- [Background] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Background] Foulks, G. N., Lemp, M., Jester, J., Sutphin, J., Murube, J., & Novack, G. (2007). report of the international dry eye workshop (DEWS). Ocul Surf, 5(2), 65-204. Foulks, G. N., Lemp, M., Jester, J., Sutphin, J., Murube, J., & Novack, G. (2007). Report of the international dry eye workshop (DEWS). Ocul Surf, 5(2), 65-204.
- [Background] Geerling G, Tauber J, Baudouin C, Goto E, Matsumoto Y, O'Brien T, Rolando M, Tsubota K, Nichols KK. The international workshop on meibomian gland dysfunction: report of the subcommittee on management and treatment of meibomian gland dysfunction. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):2050-64. doi: 10.1167/iovs.10-6997g. No abstract available. PMID 21450919
- [Background] Hom M, De Land P. Prevalence and severity of symptomatic dry eyes in Hispanics. Optom Vis Sci. 2005 Mar;82(3):206-8. doi: 10.1097/01.opx.0000156310.45736.fa. PMID 15767875
- [Background] Johnson ME, Murphy PJ. Changes in the tear film and ocular surface from dry eye syndrome. Prog Retin Eye Res. 2004 Jul;23(4):449-74. doi: 10.1016/j.preteyeres.2004.04.003. PMID 15219877
- [Background] Jones L, Downie LE, Korb D, Benitez-Del-Castillo JM, Dana R, Deng SX, Dong PN, Geerling G, Hida RY, Liu Y, Seo KY, Tauber J, Wakamatsu TH, Xu J, Wolffsohn JS, Craig JP. TFOS DEWS II Management and Therapy Report. Ocul Surf. 2017 Jul;15(3):575-628. doi: 10.1016/j.jtos.2017.05.006. Epub 2017 Jul 20. PMID 28736343
- [Background] Kenrick CJ, Alloo SS. The Limitation of Applying Heat to the External Lid Surface: A Case of Recalcitrant Meibomian Gland Dysfunction. Case Rep Ophthalmol. 2017 Jan 16;8(1):7-12. doi: 10.1159/000455087. eCollection 2017 Jan-Apr. PMID 28203190
- [Background] Lemp MA, Crews LA, Bron AJ, Foulks GN, Sullivan BD. Distribution of aqueous-deficient and evaporative dry eye in a clinic-based patient cohort: a retrospective study. Cornea. 2012 May;31(5):472-8. doi: 10.1097/ICO.0b013e318225415a. PMID 22378109
- [Background] Mori A, Shimazaki J, Shimmura S, Fujishima H, Oguchi Y, Tsubota K. Disposable eyelid-warming device for the treatment of meibomian gland dysfunction. Jpn J Ophthalmol. 2003 Nov-Dec;47(6):578-86. doi: 10.1016/s0021-5155(03)00142-4. PMID 14636848
- [Background] Nelson JD, Shimazaki J, Benitez-del-Castillo JM, Craig JP, McCulley JP, Den S, Foulks GN. The international workshop on meibomian gland dysfunction: report of the definition and classification subcommittee. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1930-7. doi: 10.1167/iovs.10-6997b. Print 2011 Mar. No abstract available. PMID 21450914
- [Background] Pult H, Riede-Pult BH, Purslow C. A comparison of an eyelid-warming device to traditional compress therapy. Optom Vis Sci. 2012 Jul;89(7):E1035-41. doi: 10.1097/OPX.0b013e31825c3479. PMID 22729167
- [Background] Qiao J, Yan X. Emerging treatment options for meibomian gland dysfunction. Clin Ophthalmol. 2013;7:1797-803. doi: 10.2147/OPTH.S33182. Epub 2013 Sep 9. PMID 24043929
- [Background] Schaumberg DA, Nichols JJ, Papas EB, Tong L, Uchino M, Nichols KK. The international workshop on meibomian gland dysfunction: report of the subcommittee on the epidemiology of, and associated risk factors for, MGD. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1994-2005. doi: 10.1167/iovs.10-6997e. Print 2011 Mar. No abstract available. PMID 21450917
- [Background] Wang MT, Jaitley Z, Lord SM, Craig JP. Comparison of Self-applied Heat Therapy for Meibomian Gland Dysfunction. Optom Vis Sci. 2015 Sep;92(9):e321-6. doi: 10.1097/OPX.0000000000000601. PMID 25955642
- [Background] Wang X, Lu X, Yang J, Wei R, Yang L, Zhao S, Wang X. Evaluation of Dry Eye and Meibomian Gland Dysfunction in Teenagers with Myopia through Noninvasive Keratograph. J Ophthalmol. 2016;2016:6761206. doi: 10.1155/2016/6761206. Epub 2016 Jan 6. PMID 26881059
- [Background] Stetson G. & Kenrick Ch. (2018). A comparision of four warm compress devices. The Association of Research in Vision and Ophthalmology (ARVO). Honolulu Hawaii. 953-B0131.